CLINICAL TRIAL: NCT05917002
Title: MPFC Theta Burst Stimulation as a Tool to Affect Rational Decision Making
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trainee Investigator did not come to institution.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro00126644
Record Dates: First submitted 2023-03-29; First posted 2023-06-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive active or sham stimulation either first or second. All participants will receive active and sham during the study, only the order will be randomized.
Who Masked: Participant, Investigator
Masking Description: This study is double blinded. Both the investigators and the participants will be blinded as to which method of stimulation they receive first.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real TBS to the mPFC (Experimental): The type of stimulation to be used will be intermittent theta burst (iTBS) stimulation to the mPFC with a figure 8 coil (Coil Cool-B65 A/P). Participants will receive three 3-minute sessions of iTBS (600 pulses; 190s; 120% resting motor threshold) with 10-15-minute breaks in between each session or more per participant preference.
  Interventions: Device: Real TBS to mPFC
- Sham TBS to the mPFC (Sham Comparator): The MagVenture MagPro system has an integrated, active sham which passes current through two surface electrodes placed on the scalp. The electrodes will be placed on the left frontalis muscle for all sessions. A patient identification card will randomize participants to receive either sham or active stimulation in the first session.This system maintains blinding by a gyroscope in the coil which indicates to the clinical staff whether the coil should be rotated up or down for this participant once the card is entered into the machine. One side of the coil is active, the other is sham. The integrity of the double blind procedure will be assessed by asking the patients and study personnel rate their confidence regarding whether they thought they received real or sham. (Scale 1-10)
  Interventions: Device: Sham TBS to mPFC

INTERVENTIONS:
Device: Real TBS to mPFC — This will be delivered with the Magventure MagPro System; (double blinded using the integrated active sham system).
  Arms: Real TBS to the mPFC
Device: Sham TBS to mPFC — This will be delivered with the Magventure MagPro System; (double blinded using the integrated active sham system). The Magventure MagPro system has an integrated active sham that passes current through two surface electrodes placed on the scalp. The electrodes are placed on the left frontalis muscle under the coil for both the real and sham stimulation sessions.
  Arms: Sham TBS to the mPFC

SUMMARY:
This is a study to investigate if a device that temporarily changes brain activity (repetitive transcranial magnetic stimulation, rTMS) might be used to change how healthy participants make decisions. This study involves 2 visits to MUSC that will each take between 2-3 hours. This study is not a treatment study, but it could help inform studies investigating treatment in the future. Participants in this study will be compensated for their time.

DETAILED DESCRIPTION:
This study aims to investigate whether a single session of excitatory repetitive transcranial magnetic stimulation (rTMS) compared to electrical sham stimulation to the medial prefrontal cortex (mPFC) facilitates rational decision making. Our prior data suggests that decisions are biased depending on if the available options are presented with a negative or positive connotation (even in the case of mathematical equivalence). Work by us and others has demonstrated that even if both options are equal, the negatively framed choice is most often avoided.

ELIGIBILITY:
Inclusion Criteria:

* Is able to read consent document and provide informed consent
* English is first or primary language

Exclusion Criteria:

* • Current psychiatric disorder (as defined by DSM-5 and determined using standardized self-report instruments)

  * Suicide attempt in the past year
  * Lifetime diagnosis of psychotic disorder or bipolar mania
  * Presence of neurological disorder that contraindicates TMS or neurophysiological recording:
  * Seizure disorder
  * Lifetime history of traumatic brain injury with loss of consciousness
  * Neurodegenerative disorder (e.g., Alzheimer's Disease, Parkinson's Disease, Frontotemporal Dementia)
  * Presence of standard contraindications for rTMS
  * Currently pregnant
  * Significant sensitivity to noise
  * Medical treatments or conditions that lower seizure threshold
  * History of severe brain injury
  * History of seizures/epilepsy
  * Currently taking chronic opiate medications or substances
  * Inability or unwillingness of subject to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Baratt Impulsiveness Scale | Change assessed at visit 1 (day 1) and visit 2 (day 2)
  Change in 30-item self-report scale that is commonly used to measure impulsiveness. Participants respond to each item using a 4-point Likert scale: 1 (rarely/never), 2 (occasionally), 3 (often), and 4 (almost always/always).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McTeague, Ph.D., Principal Investigator — Medical University of South Carolina